CLINICAL TRIAL: NCT00830154
Title: A 3 Arm, Double-blind, Placebo-controlled Parallel Group Study to Assess the Efficacy,Safety and Tolerability of Pagoclone for Adults With Stuttering
Brief Title: A Study to Assess the Efficacy and Safety of Pagoclone for Adults With Stuttering
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IP456-041
Record Dates: First submitted 2009-01-25; First posted 2009-01-27 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Stuttering
Keywords: stutter; stuttering; Adults with a history of stuttering
MeSH Terms: conditions — Stuttering | interventions — pagoclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 0.30 mg pagoclone BID
  Interventions: Drug: pagoclone
- 2 (Experimental): 0.60 mg pagoclone BID
  Interventions: Drug: pagoclone
- 3 (Placebo Comparator): placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: pagoclone — 0.30 mg BID, 0.60 mg BID
  Arms: 1; 2
Other: placebo — placebo
  Arms: 3

SUMMARY:
A multicenter, randomized, 3 arm, placebo-controlled clinical trial to assess the efficacy, safety and tolerability of pagoclone for adults with stuttering.

DETAILED DESCRIPTION:
A multicenter, randomized, 3-arm, placebo controlled, parallel group study with 24 weeks of double blind treatment followed by an 8 week double blind washout and then long-term open-label extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Male and females age 18 to 80 years presenting with a history of stuttering with onset prior to age 8 years old.
* Stuttering severity must be notable for > 3 syllables stuttered on a reading and cenversational task at scereening and with at least 2% contributed individually from conversational and reading tasks.

Exclusion Criteria:

* Patients with unstable hematological, autoimmune, endocrine, neurological, renal, hepatic, retinal, gastrointestinal, or cardiovascular disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To assess whether treatment with pagoclone 0.30 mg BID or 0.60 mg BID reduces the percentage of syllables stuttered in people who stutter compared with placebo. | Weeks 8, 16 and 24

SECONDARY OUTCOMES:
Improvement in the Clincal Global Impressions-improvement (CGI-I)scale. Patient Global Assessment of Stuttering (PGS-S) assessment. Liebowitz Social Anxiety Scale (LSAS) scores. | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Indianapolis, Indiana, United States

REFERENCES:
- See also: Click here for more information about this study — http://www.stutteringstudy.com